CLINICAL TRIAL: NCT06092073
Title: Efficacy and Safety of Bilateral Recto-Intercostal Fascial Plane Block on Perioperative Analgesia in Epigastric Hernia Repair : A Randomized Controlled Trial
Brief Title: Bilateral Recto-Intercostal Fascial Plane Block in Epigastric Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR330/9/23
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Recto-intercostal Fascial Plane Block; Epigastric Hernia; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIFPB group (Experimental): Patients will receive bilateral Recto-Intercostal Fascial Plane Block (RIFPB) using 20 mL of bupivacaine 0.25% on each side.
  Interventions: Procedure: recto-intercostal fascial plane block; Drug: bupivacaine
- Control group (No Intervention): Patients will not receive the block.

INTERVENTIONS:
Procedure: recto-intercostal fascial plane block — Patients will receive bilateral recto-intercostal fascial plane block using 20 mL of bupivacaine 0.25% on each side.
  Arms: RIFPB group
Drug: bupivacaine — bupivacaine 0.25%
  Arms: RIFPB group

SUMMARY:
The aim of this study is to evaluate the efficacy and safety bilateral recto-intercostal fascial plane block (RIFPB) in epigastric hernia.

DETAILED DESCRIPTION:
Epigastric hernias are usually occult in obese patients, and their symptoms may mimic peptic ulcer or gallbladder disease . Hernia repair is associated with considerable postoperative pain.

The recto-intercostal fascial plane block (RIFPB) is a new novel approach that was developed by Tulgar et al., 2023 who hypothesized that when we inject a local anesthetic into the interfacial plane just inferolateral to the xiphoid, between the rectus abdominis muscle and the 6-7th costal cartilages (hence, between the cartilages and the intercostal muscles between them), blockade of the anterior branches of the nerves passing through this area can be guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for elective epigastric hernia repair.

Exclusion Criteria:

* Obese patients with body mass index (BMI) >35 kg/m2.
* Patients with a large hernia containing bowel.
* Patients with local anesthetic allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-21 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Rescue analgesia in the form of 3 mg of IV morphine will be given if the numeric rating scale (NRS) score > 3. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").

SECONDARY OUTCOMES:
Total morphine consumption in the 1st 24hr | 24 hours postoperatively
  Rescue analgesia in the form of 3 mg of IV morphine will be given if the numeric rating scale (NRS) score> 3.
Pain score | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Numeric Rating Scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").
  Postoperative pain using NRS at rest and during coughing or movement will be measured at PACU, 2h. 4hr, 6h, 8h, 12h, 18h and 24h postoperative
Intraoperative fentanyl consumption | Intraoperatively.
  Additional bolus doses of fentanyl 1 µg/kg IV will be given if there is increase in heart rate or mean arterial blood pressure more than 20% of the base line (after exclusion of other causes than pain).
Intraoperative mean arterial pressure | Till the end of surgery.
  Mean arterial pressure (MAP) will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Intraoperative heart rate | Till the end of surgery.
  Heart rate (HR) will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Complications | 24 hours postoperatively
  Such as pneumothorax, nausea, vomiting, hematoma, hypotension, bradycardia and local anesthetic toxicity will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.